CLINICAL TRIAL: NCT05363384
Title: A Randomized, Open, Single-dose, Crossover-design, Phase I Study to Evaluate Bioequivalence After Co-administration of ALO 25 mg and MET XR 1,000 mg or Administration of CT-L01 25/1,000 mg in Healthy Volunteers
Brief Title: A Bioequivalence Study of CT-L01 Compared to Co-administration (ALO 25 mg and MET XR 1,000 mg) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CT-L01-101
Record Dates: First submitted 2022-04-19; First posted 2022-05-05 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-L01 25/1,000 mg FDC Tablet (Experimental): Alogliptin Benzoate 25 mg/Metformin HCl XR 1,000 mg, FDC Tablet
  Interventions: Drug: CT-L01
- Alogliptin Benzoate 25 mg, Metformin HCl XR 1,000 mg (Active Comparator): 1. Alogliptin Benzoate 25 mg
  2. Metformin HCl XR 1,000 mg
  Interventions: Drug: Alogliptin Benzoate 25 mg; Drug: Metformin HCl XR 1,000 mg

INTERVENTIONS:
Drug: CT-L01 — FDC tablet, single dose, oral administration
  Arms: CT-L01 25/1,000 mg FDC Tablet
Drug: Alogliptin Benzoate 25 mg — Alogliptin Benzoate 25 mg, oral administration
  Arms: Alogliptin Benzoate 25 mg, Metformin HCl XR 1,000 mg
Drug: Metformin HCl XR 1,000 mg — Metformin HCl XR 1,000 mg, oral administration
  Arms: Alogliptin Benzoate 25 mg, Metformin HCl XR 1,000 mg

SUMMARY:
This is a randomized, open, single-dose, crossover-design, phase 1, single-center study to evaluate bioequivalence after co-administration of ALO and MET XR or administration of CT-L01 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject aged 19 to 50 years, at screening
* A subject who weighs 50 kg or more at the screening visit and has a body mass index (BMI) of 18.0~30.0 kg/m2
* A subject who is judged to be eligible to participate by the results of screening tests (vital signs, clinical laboratory tests, 12-lead ECG, etc.) by the principal investigator within 28 days before the first administration of the investigational drug
* A subject and their partner who agree to use a medically appropriate method of contraception to exclude potential of pregnancy and not to provide sperm or ova from the first dose to 28 days after the last dose of the investigational drug
* A subject who voluntarily signs the consent form after hearing and understanding the purpose and content of this study, thge characteristics of the investigational drugs, expected adverse reactions, and etc.

Exclusion Criteria:

* A subject who has a history or present symptoms of clinically significant liver, kidney, nervous system, respiratory system, digestive system, endocrine system, blood/tumor, urinary system, cardiovascular system, musculoskeletal disease, or psychiatric disease
* A subject who has an acute illness within 28 days prior to the first dose of investigational drug
* A subject who has a history of gastrointestinal surgery that may affect drug absorption (except simple appendectomy or hernia surgery) or has gastrointestinal diseases
* A subject who has taken drugs that induce or inhibit drug metabolizing enzymes such as barbiturates within 1 month prior to the first administration
* A subject who has participated in other clinical trials or bioequivalence studies within 6 months prior to the first dose of the investigational drug
* A subject who is judged unsuitable to participate in this study by the principal investigator

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-06-11 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
AUClast (Area under the plasma concentration-time curve) | Pre-dose(0.00), 0.25, 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00, and 72.00 hours
Cmax (Peak Plasma Concentration) | Pre-dose(0.00), 0.25, 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00, and 72.00 hours

SECONDARY OUTCOMES:
AUCinf (Area under the plasma concentration-time curve from time 0 to infinity) | Pre-dose(0), 0.25, 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00, and 72.00 hours
AUClast/AUCinf | Pre-dose(0), 0.25, 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00, and 72.00 hours
Tmax (Time of peak plasma concentration) | Pre-dose(0), 0.25, 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00, and 72.00 hours
t1/2 (Half-life) | Pre-dose(0), 0.25, 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00, and 72.00 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea